CLINICAL TRIAL: NCT04100837
Title: Effect of Multiple Instrumentation in Transportal and Transtibial Techniques for ACL Reconstruction Regarding Bacterial Contamination: A Randomized Control Study
Brief Title: Multiple Instrumentation for ACL Reconstruction Regarding Bacterial Contamination
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerollos Zaghloul Thabet, Orthopedics & traumatology doctor, Assiut University
Other Study IDs: contamination of ACL surgery
Record Dates: First submitted 2019-09-14; First posted 2019-09-24 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — After preparation, swabs will be obtained from subcutaneous tissue at antromedial portal track in transportal technique (femoral tunnel drilling) and in transtibial technique before and after the instrumentation and femoral screw insertion, a control sample will be taken at antrolateral track in both techniques, then samples will be sended to the lab to be studied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transportal group: swabs will be obtained from subcutaneous tissue at antromedial portal track in transportal technique (femoral tunnel drilling) , before and after the instrumentation and femoral screw insertion, a control sample will be taken at antrolateral track in both techniques, then samples will be sended to the lab to be studied.
- transtibial group: swabs will be obtained from subcutaneous tissue at antromedial portal track in transtibial technique (femoral tunnel drilling), before and after the instrumentation and femoral screw insertion, a control sample will be taken at antrolateral track in both techniques, then samples will be sended to the lab to be studied.

SUMMARY:
To determine the Effect of multiple instrumentation regarding bacterial contamination in transportal and transtibial techniques in ACL reconstruction .A Randomized controlled study

DETAILED DESCRIPTION:
Infection is a catastrophic and one of the most dreaded complications in orthopaedic surgery. Several measures have been undertaken to reduce the risk of infection, one of which is the use of systemic prophylactic antibiotics.

The purpose of this study is to determine the effect of multiple instrumentation regarding bacterial contamination in transportal and transtibial techniques in ACL reconstruction . About Eighty consecutive patients having surgical indication for ACL-R will be included, the cases will be divided into two groups, 35 cases will undergo for the transtibial technique and the other 45 cases will undergo for the transportal technique. After preparation, swabs will be obtained from subcutaneous tissue at antromedial portal track in transportal technique (femoral tunnel drilling) and in transtibial technique before and after the instrumentation and femoral screw insertion, a control sample will be taken at antrolateral track in both techniques, then samples will be sended to the lab to be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated ACL Injury.
2. Non deformed knee.

Exclusion Criteria:

1. Associated knee injury (eg. PCL).
2. Deformed knee ( eg. genu varus , genu valgus more than 4 degree )
3. patient with medical history of being immune compromized patient eg,DM

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Total coverage of all eligible cases will be admitted to Arthoscopic Unit within 6 months
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Assessment the concentration of contamination in ACL operation. | Through study completion, an average of 1 year.
  Effect of instrumentation on contamination of the operation,swabs will be obtained intraoperative for cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham HK El-kadi, professor, Study Director — Assiut University
Locations (1):
- Assiut Univeristy, Asyut, Egypt

REFERENCES:
- [Background] Barnstable CJ, Jones EA, Bodmer WF, Bodmer JG, Arce-Gomez B, Snary D, Crumpton MJ. Genetics and serology of HL-A-linked human Ia antigens. Cold Spring Harb Symp Quant Biol. 1977;41 Pt 2:443-55. doi: 10.1101/sqb.1977.041.01.052. No abstract available. PMID 70300